CLINICAL TRIAL: NCT03406208
Title: Resiliency Training for Adults With Neurofibromatosis Via Live Videoconferencing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Clinical Psychologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017P000143; W81XWH-17-1-0121 (Other Grant/Funding Number: United States Department of Defense)
Record Dates: First submitted 2017-12-06; First posted 2018-01-23 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Neurofibromatoses; Neurofibromatosis 1; Neurofibromatosis 2; Schwannomatosis
Keywords: Psychiatry; Psychology; Psychosocial; Behavioral
MeSH Terms: conditions — Neurofibromatoses; Neurofibromatosis 1; Neurofibromatosis 2; Schwannomatosis; Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress and Symptom Management Program 1 (Experimental): The Stress and Symptom Management Program 1 (SMP1) introduces and reinforces stress and symptom management skills. The program consists of 8 weekly sessions (90 minutes each), delivered through live videoconferencing.
  Interventions: Behavioral: Stress and Symptom Management Program 1
- Stress and Symptom Management Program 2 (Experimental): The Stress and Symptom Management Program 2 (SMP2) introduces and reinforces stress and symptom management skills. The program consists of 8 weekly sessions (90 minutes each), delivered through live videoconferencing.
  Interventions: Behavioral: Stress and Symptom Management Program 2

INTERVENTIONS:
Behavioral: Stress and Symptom Management Program 1 — The Stress and Symptom Management Program 1 (SMP1) introduces and reinforces stress and symptom management skills. The program consists of 8 weekly sessions (90 minutes each), delivered through live videoconferencing.
  Other Names: SMP2
  Arms: Stress and Symptom Management Program 1
Behavioral: Stress and Symptom Management Program 2 — The Stress and Symptom Management Program 2 (SMP2) introduces and reinforces stress and symptom management skills. The program consists of 8 weekly sessions (90 minutes each), delivered through live videoconferencing.
  Other Names: SMP2
  Arms: Stress and Symptom Management Program 2

SUMMARY:
The aims of this study are to compare the effect and durability of two stress and symptom management programs tailored for patients with neurofibromatosis on quality of life and psychosocial functioning.

DETAILED DESCRIPTION:
The aims of this study are to compare the effect of two stress and symptom management programs tailored for patients with neurofibromatosis on quality of life and psychosocial functioning. We will also examine the degree to which treatment-dependent improvements in quality of life are mediated by improvements in depression, anxiety, distress, mindfulness, gratitude, social support, empathy, optimism, coping, pain intensity and pain interference.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of NF1, NF2, or Schwannomatosis
* 18 years of age or older
* Is capable of completing and fully understanding the informed consent process, study procedures, and study assessments in English
* At least 6th grade self-reported reading level
* Self-reported difficulties coping with stress and NF-symptoms
* Score of 6 or higher on Perceived Stress Scale 4-Item (PSS-4)

Exclusion Criteria:

* Has major medical comorbidity not NF related expected to worsen in the next 12 months
* Recent (within past 3 months) change in antidepressant medication
* Recent (within past 3 months) participation in cognitive behavioral therapy or relaxation therapy
* Has significant mental health diagnosis requiring immediate treatment (e.g., bipolar disorder, psychotic disorder, active substance use dependence)
* Unable or unwilling to complete assessments electronically via REDCap
* Unable or unwilling to participate in group videoconferencing sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Physical Quality of Life | 0 Weeks, 8 Weeks, 6 Months, 12 Months
  World Health Organization Quality of Life Brief (WHOQOL-BREF); 4-20; higher score indicates higher QoL
Change in Psychological Quality of Life | 0 Weeks, 8 Weeks, 6 Months, 12 Months
  World Health Organization Quality of Life Brief (WHOQOL-BREF); 4-20; higher score indicates higher QoL

SECONDARY OUTCOMES:
Social Quality of Life | 0 Weeks, 8 Weeks, 6 Months, 12 Months
  World Health Organization Quality of Life Brief (WHOQOL-BREF); 4-20; higher score indicates higher QoL
Environmental Quality of Life | 0 Weeks, 8 Weeks, 6 Months, 12 Months
  World Health Organization Quality of Life Brief (WHOQOL-BREF); 4-20; higher score indicates higher QoL
Depression | 0 Weeks, 8 Weeks, 6 Months, 12 Months
  Patient Health Questionnaire 9-Item (PHQ-9); 0-27; higher score indicates more symptoms of depression
Anxiety | 0 Weeks, 8 Weeks, 6 Months, 12 Months
  Generalized Anxiety Disorder 7-Item (GAD-7); 0-21; higher score indicates more symptoms of anxiety
Social Support | 0 Weeks, 8 Weeks, 6 Months, 12 Months
  Medical Outcome Study Social Support Survey (MOS); 18-90; higher scores indicate greater perceived social support
Gratitude | 0 Weeks, 8 Weeks, 6 Months, 12 Months
  Gratitude Questionnaire 6-Item (GQ-6); 6-42; higher scores indicate greater gratitude
Optimism | 0 Weeks, 8 Weeks, 6 Months, 12 Months
  Life Orientation Test-Revised (LOT-R); 0-40; higher scores indicate greater optimism
Coping Strategies | 0 Weeks, 8 Weeks, 6 Months, 12 Months
  Measure of Current Status Part A (MOCS-A); 0-52; higher scores indicate greater perceived ability to cope
Mindfulness | 0 Weeks, 8 Weeks, 6 Months, 12 Months
  Cognitive and Affective Mindfulness Scale (CAMS); 10-40; higher scores indicate greater mindfulness
Empathy | 0 Weeks, 8 Weeks, 6 Months, 12 Months
  Interpersonal Reactivity Index (IRI) Empathy Subscale; 7-Items; 0-28; higher scores indicate greater empathy
Pain Intensity | 0 Weeks, 8 Weeks, 6 Months, 12 Months
  Graded Chronic Pain Scale (GCPS); 0-100; higher scores indicate greater pain intensity
Pain Interference | 0 Weeks, 8 Weeks, 6 Months, 12 Months
  PROMIS Pain Interference; 8-40; higher scores indicate more pain interference
Stress | 0 Weeks, 8 Weeks, 6 Months, 12 Months
  Perceived Stress Scale 10-Item (PSS-10); 0-21; higher scores indicate greater levels of perceived stress

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Maria Vranceanu, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brewer JR, Hooker JE, Kanaya M, LaCamera DE, Bakhshaie J, Vranceanu AM. Social support moderates quality of life outcomes during a mind-body intervention among adults with neurofibromatosis. J Neurooncol. 2025 Oct;175(1):133-141. doi: 10.1007/s11060-025-05108-8. Epub 2025 Aug 7. PMID 40773151
- [Derived] Hooker JE, Doorley JD, Greenberg J, Bakhshaie J, Manglani HR, Briskin EA, Vranceanu AM. Improvements in pain interference among geographically diverse adults with neurofibromatosis: Results from a fully powered randomized controlled trial. Neurooncol Pract. 2024 Sep 20;12(1):58-67. doi: 10.1093/nop/npae084. eCollection 2025 Feb. PMID 39917761
- [Derived] McDermott K, Bakhshaie J, Brewer J, Vranceanu AM. The impact of a virtual mind-body program on symptoms of depression and anxiety among international English-speaking adults with neurofibromatosis. Am J Med Genet A. 2024 Jun;194(6):e63543. doi: 10.1002/ajmg.a.63543. Epub 2024 Feb 6. PMID 38318960
- [Derived] Presciutti AM, Lester EG, Woodworth EC, Greenberg J, Bakhshaie J, Hooker JE, McDermott KA, Vranceanu AM. The impact of a virtual mind-body program on resilience factors among international English-speaking adults with neurofibromatoses: secondary analysis of a randomized clinical trial. J Neurooncol. 2023 Jul;163(3):707-716. doi: 10.1007/s11060-023-04389-1. Epub 2023 Jul 13. PMID 37440099
- [Derived] Vranceanu AM, Manglani HR, Choukas NR, Kanaya MR, Lester E, Zale EL, Plotkin SR, Jordan J, Macklin E, Bakhshaie J. Effect of Mind-Body Skills Training on Quality of Life for Geographically Diverse Adults With Neurofibromatosis: A Fully Remote Randomized Clinical Trial. JAMA Netw Open. 2023 Jun 1;6(6):e2320599. doi: 10.1001/jamanetworkopen.2023.20599. PMID 37378983
- [Derived] Lester EG, Wang KE, Blakeley JO, Vranceanu AM. Occurrence and Severity of Suicidal Ideation in Adults With Neurofibromatosis Participating in a Mind-Body RCT. Cogn Behav Neurol. 2023 Mar 1;36(1):19-27. doi: 10.1097/WNN.0000000000000332. PMID 36651958
- [Derived] Fishbein NS, Vranceanu AM, Mace RA. Baseline characteristics of adults with neurofibromatosis enrolled on a psychosocial randomized controlled trial. J Neurooncol. 2022 Sep;159(3):637-646. doi: 10.1007/s11060-022-04104-6. Epub 2022 Aug 4. PMID 35925531
- [Derived] Bannon SM, Hopkins SW, Grunberg VA, Vranceanu AM. Psychosocial profiles of risk and resiliency in neurofibromatoses: a person-centered analysis of illness adaptation. J Neurooncol. 2022 Feb;156(3):519-527. doi: 10.1007/s11060-021-03928-y. Epub 2022 Jan 22. PMID 35064449
- [Derived] Mace RA, Doorley J, Bakhshaie J, Cohen JE, Vranceanu AM. Psychological resiliency explains the relationship between emotional distress and quality of life in neurofibromatosis. J Neurooncol. 2021 Nov;155(2):125-132. doi: 10.1007/s11060-021-03852-1. Epub 2021 Sep 27. PMID 34570301
- [Derived] Doorley JD, Greenberg J, Bakhshaie J, Fishbein NS, Vranceanu AM. Depression explains the association between pain intensity and pain interference among adults with neurofibromatosis. J Neurooncol. 2021 Sep;154(2):257-263. doi: 10.1007/s11060-021-03826-3. Epub 2021 Aug 19. PMID 34409538
- [Derived] Lester EG, Gates MV, Vranceanu AM. Mind-Body Therapy via Videoconferencing in Patients With Neurofibromatosis: Analyses of 1-Year Follow-up. Ann Behav Med. 2021 Feb 12;55(1):77-81. doi: 10.1093/abm/kaaa030. PMID 32421171
- [Derived] Vranceanu AM, Zale EL, Funes CJ, Macklin EA, McCurley J, Park ER, Jordan JT, Lin A, Plotkin SR. Mind-Body Treatment for International English-Speaking Adults With Neurofibromatosis via Live Videoconferencing: Protocol for a Single-Blind Randomized Controlled Trial. JMIR Res Protoc. 2018 Oct 23;7(10):e11008. doi: 10.2196/11008. PMID 30355560